CLINICAL TRIAL: NCT05476432
Title: Hepatic Arterial Infusion With Oxaliplatin & 23h Fluorouracil Versus Hepatic Arterial Infusion With Oxaliplatin & 46h Fluorouracil for Unresectable Hepatocellular Carcinoma：a Non-inferiority Study
Brief Title: HAIC With One-day FOLFOX vs. HAIC With Two-day FOLFOX for Unresectable HCC: a Non-inferiority Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou No.12 People's Hospital (Other Government); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH-5
Record Dates: First submitted 2022-07-26; First posted 2022-07-27 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC 1d (Experimental): Oxaliplatin, leucovorin, and bolus fluorouracil were conducted equally in the both groups, while infusional fluorouracil 2400 mg/m² was given over 23 hours in the HAIC 1d group
  Interventions: Procedure: HAIC; Drug: FOLFOX 1d
- HAIC 2d (Active Comparator): Oxaliplatin, leucovorin, and bolus fluorouracil were conducted equally in the both groups, while infusional fluorouracil 2400 mg/m² was given over 46 hours in the HAIC 2d group
  Interventions: Procedure: HAIC; Drug: FOLFOX 2d

INTERVENTIONS:
Procedure: HAIC — The microcatheter was advanced into the hepatic artery, and patients were transferred to the inpatient ward for drug infusion via the hepatic artery
Drug: FOLFOX 2d — Oxaliplatin, leucovorin, bolus fluorouracil, and infusional fluorouracil 2400 mg/m² over 46 hours
  Arms: HAIC 2d
Drug: FOLFOX 1d — Oxaliplatin, leucovorin, bolus fluorouracil, and infusional fluorouracil 2400 mg/m² over 23 hours
  Arms: HAIC 1d

SUMMARY:
Hepatic arterial infusion chemotherapy (HAIC) with oxaliplatin&5-fluorouracil was effective in unresectable hepatocellular carcinoma (HCC). The program of FOLFOX-HAIC in HCC was performed for 1 day (HAIC 1d) or 2 days (HAIC 2d). We hereby retrospectively compared the efficacy and safety between these two treatment regimens, and explored the predictive power of thymidylate synthase (TYMS), an enzyme involved in the DNA synthesis process and metabolism of fluorouracil. Patients with HCC staged BCLC A-B receive HAIC only, and patients with HCC staged BCLC C receive HAIC plus systemic treatment, such as sorafenib, A+T, lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18-75 years;
* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL), simultaneously staged as BCLC A, BCLC B or BCLC C based on Barcelona Clinic Liver Cancer staging system.
* Patients must have at least one tumor lesion that can be accurately measured
* Diagnosed as unresectable with consensus by the panel of liver surgery experts
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* Poor compliance that can not comply with the course of treatment and follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  time from randomzation to death

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  time from randomzation to progression or death, which occur firstly.
objective response rate per RECIST 1.1 | 12 months
  CR plus PR per RECIST 1.1
Adverse Events | 30 days
  Adverse Events according to CTCAE 4.0
the predictive power of thymidylate synthase (TYMS) | 12 months
  the correlation between thymidylate synthase (TYMS) and survival. Whether the survival of patients with low TYMS is better than those with high TYMS

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong